CLINICAL TRIAL: NCT03477968
Title: ThRombosis ExclUsion STudy
Acronym: TRUST
Status: Terminated | Type: Observational
Why Stopped: Due to the unstability of samples included in the plasmabank using the reference method: VIDAS system, Stago decided to not use the plasmabank to assess the pre-specified primary objective. Therefore, this study was halted prematurely.
Sponsor: Diagnostica Stago (Industry)
Responsible Party: Sponsor
Other Study IDs: TRUST study
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Deep Venous Thromboses; Pulmonary Embolism; Venous Thromboembolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pulmonary Embolism (PE): Patients presenting with PE suspicion. Diagnosis will be performed according to Standard of Care. Plasma samples will be collected if PTP score is Low or Moderate. If diagnosis is negative, patients will be followed for 3 months to evaluate potential VTE development.
  Enrolment completed for this group : 13th February 2020
  Interventions: Diagnostic Test: DDimer test
- Deep Venous Thrombosis (DVT): Patients presenting with DVT suspicion. Diagnosis will be performed according to Standard of Care. Plasma samples will be collected if PTP score is Low or Moderate. If diagnosis is negative, patients will be followed for 3 months to evaluate potential VTE development.
  Enrolment completed for this group : 29th March 2023
  Interventions: Diagnostic Test: DDimer test

INTERVENTIONS:
Diagnostic Test: DDimer test — Measuring the level of DDimer in blood sample

SUMMARY:
Primary objective: To demonstrate the ability of STA® - Liatest® D-Di XL combined with a clinical PreTest Probability (PTP) to safely exclude pulmonary embolism (PE) and deep venous thrombosis (DVT) as measured by Negative Predictive Value (NPV) and sensitivity.

Secondary objectives:

1. To estimate additional STA® - Liatest® D-Di XL accuracy parameters, including specificity and positive predictive value (PPV)
2. To constitute a plasma bank to be used for future studies with other DDi assays under development by Stago.

DETAILED DESCRIPTION:
The study population will be selected from prospective, consecutive ambulatory outpatients suspected of having venous thromboembolism. Patients will be diagnosed for VTE (PE or DVT) based on local standard of care. Samples will be collected (additional blood draw or additional volume during blood draw) for future testing with new D-Dimer assay.

In case of Low/Moderate PTP score and negative VTE diagnosis, patients will be followed for 3 months to evaluate potential development of deep venous thrombosis and/or pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is < 80 years old.
2. Patient presents at least one of these symptoms indicative of proximal DVT or PE:

   * symptoms for proximal DVT: leg pain, tenderness (discomfort through palpation), leg swelling, and /or edema,
   * symptoms for PE: hemoptysis, lung related chest pain, dyspnea.
3. Patient provides written informed consent to participate in the study
4. Patient is willing to comply with specified follow-up evaluation at 3 months and can be contacted by telephone.

Exclusion Criteria:

1. Patient presenting with a condition that may be associated with increased D-dimer levels, even in the absence of VTE, such as:

   * Fibrinolytic therapy within the previous seven (7) days,
   * Disseminated intravascular coagulation
   * Bone fracture or surgery (with general anesthesia longer than thirty (30) minutes) within the previous one (1) month,
   * Deep hematoma diagnosed by imaging techniques within the previous one (1) month,
   * Disseminated malignancies and active cancer (active cancer defined as: cancer for which therapeutic or palliative treatment is either ongoing at the time of enrolment or has stopped less than six (6) months before enrolment),
   * Sepsis, severe infections, pneumonia within the previous 1 month,
   * Known liver cirrhosis,
   * Pregnancy or having delivered within the previous 1 month,
   * Atherosclerotic vascular disease thrombosis within the previous 1month (e.g. myocardial infarction, stroke, coronary syndrome, peripheral artery disease stage III or IV),
   * Sickle cell disease,
2. Patients presenting with a suspect thrombotic event related to catheter implantation
3. Ongoing therapeutic anticoagulants (curative and preventive regimen) started twenty four (24) hours or more before blood draw (except aspirin and platelet inhibitors)
4. Previous anticoagulant therapy stopped less than three (3) months before blood draw (except aspirin and platelet inhibitors)
5. Patients with previous DVT/PE occurred less than three (3) months from screening.
6. Suspect thrombotic events in other locations at screening, including distal to the knee and upper extremity DVT (based on standard of care examinations)
7. Patients with known tissue plasminogen activator (tPA) deficiency
8. Patient participating or who has participated within one month of enrolment in another investigational study
9. Major co-morbid condition(s) or other reasons that could limit the patient's ability to participate in the study or to comply with follow-up requirements, or impact the scientific integrity of the study.

Max Age: 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be recruited from prospective, consecutive, ambulatory outpatients (presenting at the emergency unit or outpatient clinic) suspected of having VTE. Patients with DVT and PE will be analyzed as separate groups.
Sampling Method: Probability Sample
Enrollment: 5935 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2024-09-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (12):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Northwestern Medical Center, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - Taylor regional Hospital, Campbellsville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Duke Hemostasis and Thrombosis Research Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Lehigh Hospital, Allentown, Pennsylvania
  - St Luke's University Health Network, Bethlehem, Pennsylvania
  - Jefferson University Hospital, Philadelphia, Pennsylvania
  - UT Southwestern, Dallas, Texas
- Cliniques Universitaires St Luc, Brussels, Belgium
- France (4):
  - CHU, Angers
  - CHU, Dijon
  - CHU, Grenoble
  - CHU, Rouen
- University Hospital S. Orsola-Mapighi, Bologna, Italy
- Spain (2):
  - Hospital Universitario Virgen del Rocio, Seville
  - General Hospital, Soria

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As STA® - Liatest® D-Di XL was not available for testing before the end of the collection, it was not possible to anticipate the number of samples that might be lost during thawing due to stability. We decided to apply a 15% increase to the number of positives. Taking into account the decision to enroll N = 115 evaluable reference-positive subjects for each indication, sample size had to be recalculated. At study end, a total of 3,584 PE and 2,351 DVT subjects had been enrolled.
Groups:
- Pulmonary Embolism (PE): Patients presenting with PE suspicion. Diagnosis will be performed according to Standard of Care. Plasma samples will be collected if PTP score is Low or Moderate. If diagnosis is negative, patients will be followed for 3 months to evaluate potential VTE development.
  Enrolment completed for this group : 13th February 2020
  DDimer test: Measuring the level of DDimer in blood sample
- Deep Venous Thrombosis (DVT): Patients presenting with DVT suspicion. Diagnosis will be performed according to Standard of Care. Plasma samples will be collected if PTP score is Low or Moderate. If diagnosis is negative, patients will be followed for 3 months to evaluate potential VTE development.
Period: Overall Study
Arm/Group | Pulmonary Embolism (PE) | Deep Venous Thrombosis (DVT)
Started | 3584 | 2351
Completed | 2778 | 1622
Not Completed | 806 | 729

BASELINE CHARACTERISTICS:
Groups:
- Deep Venous Thrombosis (DVT): Patients presenting with DVT suspicion. Diagnosis will be performed according to Standard of Care. Plasma samples will be collected if PTP score is Low or Moderate. If diagnosis is negative, patients will be followed for 3 months to evaluate potential VTE development.
  Enrolment completed for this group : 29th March 2023
  DDimer test: Measuring the level of DDimer in blood sample
- Total: Total of all reporting groups
Arm/Group | Pulmonary Embolism (PE) | Deep Venous Thrombosis (DVT) | Total
Number analyzed (Participants) | 2778 | 1622 | 4400
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The primary aim of this trial was to demonstrate the ability of STA® - Liatest® D-Di XL to exclude PE and DVT in out patients with low or moderate clinical PreTest Probability for each indication separetely. In addition, during the study the enrolment in the DVT and PE arms was monitored separetely to achieve the desired sample size for each indication. Hence, this study is considered as single trial with two separate arms, the data as age were calculated only for each arm and not in total.
  years
    Pulmonary Embolism (PE) Participants: number analyzed (Participants) | 2778 | 0 | 2778
    Pulmonary Embolism (PE) Participants | 45.8 (15.2) |  | 45.8 (15.2)
    Deep Venous Thrombosis (DVT) Participants: number analyzed (Participants) | 0 | 1622 | 1622
    Deep Venous Thrombosis (DVT) Participants |  | 51.9 (14.7) | 51.9 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1675 | 994 | 2669
  Male | 1103 | 628 | 1731
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: VTE Exclusion
Description: According to the ThRombosis ExclUsion STudy (TRUST) protocol, the primary objective of the study was to demonstrate the ability of STA® - Liatest® D-Di XL combined with a clinical PreTest Probability to safely exclude pulmonary embolism (PE) and deep venous thrombosis (DVT) as measured by Negative Predictive Value (NPV) and sensitivity.
  The first step was to evaluate the stability of the plasmabank using VIDAS system. The preliminary results showed that the plasmabank was unusable with a high rate of unstable samples. Stago, decided to not use this plasmabank to assess the ability of STA® - Liatest® D-Di XL to safely exclude PE and DVT.
Time Frame: Initially, we planned to enroll subjects suspected of PE/DVT to constitute a plasmabank, then perform testing of STA- Liatest D-Di XL for on this latter on 48 months. However due to plasmabank unstability, Stago decided to not perform the testing phase.
Population: As described in the Protocol Section, the study was halted prematurely, therefore there is no Outcome Measure data.
Arm/Group | Pulmonary Embolism (PE) | Deep Venous Thrombosis (DVT)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: VTE Exclusion
Description: According to the ThRombosis ExclUsion STudy (TRUST) protocol, the secondary objectives of the study were:
  1. To estimate additional STA® - Liatest® D-Di XL accuracy parameters, including specificity and positive predictive value (PPV)
  2. To constitute a plasmabank to be used for future studies with other DDi assays under development by Stago.
  The first step was to evaluate the stability of the plasmabank using VIDAS system. The preliminary results showed that the plasmabank was unusable with a high rate of unstable samples. Stago, decided to not use this plasmabank to assess the ability of STA® - Liatest® D-Di XL to safely exclude PE and DVT and to not use this plasmabank for future studies with other DDi assays under development by Stago.
Time Frame: Initially, we planned to enroll subjects suspected of PE/DVT to constitute a plasmabank, then perform testing of STA- Liatest D-Di XL. Due to plasmabank unstability, Stago decided to not perform the testing phase for the STA-D-Di XL and future DDi assays.
Population: As described in the Protocol Section, the study was halted prematurely, therefore there is no Outcome Measure data.
Arm/Group | Pulmonary Embolism (PE) | Deep Venous Thrombosis (DVT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: In the EU / US, this was a non-interventional study in which patients received standard of care, unrelated to study procedures. As such, safety was not evaluated in this study.
Description: In the EU / US, this was a non-interventional study in which patients received standard of care, unrelated to study procedures. As such, safety was not evaluated in this study.
Groups:
- Pulmonary Embolism (PE) Arm: Patients presenting with PE suspicion. Diagnosis will be performed according to Standard of Care. Plasma samples will be collected if PTP score is Low or Moderate. If diagnosis is negative, patients will be followed for 3 months to evaluate potential VTE development.
  Enrolment completed for this group : 13th February 2020
  DDimer test: Measuring the level of DDimer in blood sample
- Deep Venous Thrombosis (DVT) Arm: Patients presenting with DVT suspicion. Diagnosis will be performed according to Standard of Care. Plasma samples will be collected if PTP score is Low or Moderate. If diagnosis is negative, patients will be followed for 3 months to evaluate potential VTE development.
  Enrolment on going : 29th March 2020
  DDimer test: Measuring the level of DDimer in blood sample
Arm/Group | Pulmonary Embolism (PE) Arm | Deep Venous Thrombosis (DVT) Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the informations regarding the PIs restrictions are specified in the study agreement for each study site.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT03477968/Prot_SAP_000.pdf